CLINICAL TRIAL: NCT03200444
Title: Evaluation of the Peel Force of New Adhesives From the Skin
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Coloplast A/S (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: CP267_01
Record Dates: First submitted 2017-06-26; First posted 2017-06-27 (Actual); Results first posted 2025-04-25 (Actual); Last update posted 2025-04-25 (Actual); Status verified 2025-04

CONDITIONS: Stoma Ileostomy
MeSH Terms: interventions — Cyclin-Dependent Kinase Inhibitor p15; Cyclin-Dependent Kinase Inhibitor p16

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Testing of 6 adhesive strips (Experimental): Each subject tests six adhesive strips on pre-striped skin.
  1. Standard adhesive 1
  2. standard adhesive 2
  3. Standard adhesive 3
  4. P-4
  5. P-15
  6. P-16
  The six strips are applied on abdominal skin. The order to which the adhesive strips are located on the skin is randomized. The subjects will change the adhesive strips at home and the adhesion of the adhesive strips will be measured at 5 visits.
  Interventions: Other: Standard adhesive 1; Other: Standard adhesive 2; Other: Standard adhesive 3; Other: P-4; Other: P-15; Other: P-16

INTERVENTIONS:
Other: Standard adhesive 1 — This strip consists of a standard hydrocolloid adhesive found in ostomy products
Other: Standard adhesive 2 — This strip consists of a standard hydrocolloid adhesive found in ostomy products
Other: Standard adhesive 3 — This strip consists of a standard hydrocolloid adhesive found in ostomy products
Other: P-4 — Newly developed adhesive P-4
Other: P-15 — Newly developed adhesive P-14
Other: P-16 — Newly developed adhesive P-8

SUMMARY:
This study investigates the impact and adhesion of new adhesives to the skin.

ELIGIBILITY:
Inclusion Criteria:

1. Have given written informed consent
2. Be at least 18 years of age and have full legal capacity
3. Have intact skin on the area used in the investigation

Exclusion Criteria:

1. Currently receiving or have within the past 2 months received radio- and/or chemotherapy
2. Currently receiving or have within the past months received topical steroid treatment in the abdominal skin area or systemic steroid (tablet/injection) treatment.
3. Are pregnant or breastfeeding
4. Have dermatological problems in the abdominal area (assessed by investigator)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2017-07-03 (Actual); Primary Completion 2020-06-30 (Actual); Study Completion 2020-06-30 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Coloplast A/S, Humlebæk, Denmark

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Units Other Than Participants: Number of strips
Groups:
- P-4 Adhesive; P-15 Adhesive; P-16 Adhesive: Newly developed adhesive
Period: Overall Study
Arm/Group | Standard Adhesive 1 | Standard Adhesive 2 | Standard Adhesive 3 | P-4 Adhesive | P-15 Adhesive | P-16 Adhesive
Started | 6; 6 Number of strips | 6; 6 Number of strips | 6; 6 Number of strips | 6; 6 Number of strips | 6; 6 Number of strips | 6; 6 Number of strips
Completed | 6; 6 Number of strips | 6; 6 Number of strips | 6; 6 Number of strips | 6; 6 Number of strips | 6; 6 Number of strips | 6; 6 Number of strips
Not Completed | 0; 0 Number of strips | 0; 0 Number of strips | 0; 0 Number of strips | 0; 0 Number of strips | 0; 0 Number of strips | 0; 0 Number of strips

BASELINE CHARACTERISTICS:
Population: Not different from the assignment in Participant Flow
Groups:
- Testing of 6 Adhesive Strips: Each subject tests six adhesive strips on pre-striped skin.
  1. Standard adhesive 1
  2. standard adhesive 2
  3. Standard adhesive 3
  4. P-4
  5. P-15
  6. P-16
  The six strips are applied on abdominal skin. The order to which the adhesive strips are located on the skin is randomized. The subjects will change the adhesive strips at home and the adhesion of the adhesive strips will be measured at 5 visits.
  Standard adhesive 1: This strip consists of a standard hydrocolloid adhesive found in ostomy products
  Standard adhesive 2: This strip consists of a standard hydrocolloid adhesive found in ostomy products
  Standard adhesive 3: This strip consists of a standard hydrocolloid adhesive found in ostomy products
  P-4: Newly developed adhesive P-4
  P-15: Newly developed adhesive P-14
  P-16: Newly developed adhesive P-8
Arm/Group | Testing of 6 Adhesive Strips
Number analyzed (Participants) | 6
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 6
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 3
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 0
  Unknown or Not Reported | 6
Region of Enrollment [Number; unit: participants]
  Denmark | 6

OUTCOME MEASURES:

1. Primary Outcome: Peel Force
Description: The peel force (N) needed to peel off adhesive strips from the skin
Time Frame: 30 min
Population: All participants were analysed
Measure: Median (Full Range); unit: Newton
Arm/Group | Standard Adhesive 1 | Standard Adhesive 2 | Standard Adhesive 3 | P-4 Adhesive | P-15 Adhesive | P-16 Adhesive
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6
Newton | 5.2 [3.3 to 5.4] | 3 [2.3 to 4.8] | 2.1 [1.6 to 4.1] | 3.3 [3.3 to 4.5] | 3.7 [2.2 to 5.0] | 4.4 [2.1 to 5.1]

ADVERSE EVENTS:
Time Frame: Adverse event data were collected over 4 weeks
Description: Any untoward or unfavorable medical occurrence in a participant, including any abnormal sign (for example, abnormal physical exam or laboratory finding), symptom, or disease, temporally associated with the participant's participation in the research, whether or not considered related to the participant's participation in the research
Arm/Group | Standard Adhesive 1 | Standard Adhesive 2 | Standard Adhesive 3 | P-4 Adhesive | P-15 Adhesive | P-16 Adhesive
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6
Other Adverse Events (participants affected / at risk) | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-06-01): https://cdn.clinicaltrials.gov/large-docs/44/NCT03200444/Prot_SAP_000.pdf